CLINICAL TRIAL: NCT06146881
Title: The Indonesian Research on Survey and Treatment for Dry Eye Disease (ThIRST DED): Effectiveness of Diquafosol Prophylactic Therapy to Prevent Dry Eye Disease for Cataract Surgery Patients in Indonesia
Brief Title: Effectiveness of Diquafosol Prophylactic Therapy to Prevent Dry Eye Disease for Cataract Surgery Patients in Indonesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Prof. Dr. dr. Ratna Sitompul, Sp.M(K), Prof. Dr. dr. Ratna Sitompul, Sp.M(K), Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21050581
Record Dates: First submitted 2023-11-09; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Disease
Keywords: Dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diquafosol sodium 3% group (Experimental): Diquafosol sodium 3% 4 times a day for 4 weeks before cataract surgery and 21 days after surgery
  Interventions: Drug: Diquafosol sodium 3%
- Sodium hyaluronate 0.1% group (Active Comparator): Sodium hyaluronate 0.1% 4 times a day for 4 weeks before cataract surgery and 21 days after surgery
  Interventions: Drug: Sodium hyaluronate 0.1%

INTERVENTIONS:
Drug: Diquafosol sodium 3% — Diquafosol sodium 3% 4 times a day for 4 weeks before cataract surgery and 21 days after surgery
  Arms: Diquafosol sodium 3% group
Drug: Sodium hyaluronate 0.1% — Sodium hyaluronate 0.1% 4 times a day for 4 weeks before cataract surgery and 21 days after surgery
  Arms: Sodium hyaluronate 0.1% group

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of preventive therapy with diquafosol sodium 3% compared to sodium hyaluronate 0.1% to prevent dry eye disease in patient who will undergo cataract surgery. The main questions it aims to answer are:

* The percentage reduction in subjective symptoms and signs of dry eye disease after cataract surgery.
* The differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs in patients objectively.
* The tear osmolarity and matix metalloproteinase-9 (MMP-9) after the treatment.
* The difference in visual quality improvement assessed from higher order aberrations (HOA) and contrast sensitivity after administration of diquafosol sodium 3% compared to sodium hyaluronate 0.1%.

Participants will receive diquafosol sodium 3% or sodium hyaluronate 0.1% for 4 weeks before the cataract surgery and 21 days after the surgery, and will be:

* Interviewed regarding their identity, history of illness, and symptoms of dry eye disease.
* Examined by researchers: eye condition, contrast sensitivity using the Pelli-Robson diagram, keratograph, HOA, tear osmolarity, MMP-9, corneal sensitivity, tear break up time (TBUT) , fluorescein break up pattern (FBUP).

This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.

DETAILED DESCRIPTION:
The general objective of this study is to determine the effectiveness of preventive therapy with diquafosol sodium 3% compared to sodium hyaluronate 0.1% for patient who will undergo cataract surgery. The objective is being measure by the reducing symptoms and milder signs of dry eye disease and improving vision quality in post-cataract surgery patients.

1. Evaluate the percentage reduction in subjective symptoms and signs of dry eye disease after cataract surgery with diquafosol sodium 3% compared to sodium hyaluronate 0.1% in patients who want to undergo cataract surgery.
2. Evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs in patients objectively by examining the value of break up time, corneal sensibility, keratograph and FBUP
3. Evaluate tear osmolarity and MMP-9 after administration of diquafosol sodium 3% compared to sodium hyaluronate 0.1%
4. Evaluate the difference in visual quality improvement assessed from HOA and contrast sensitivity after administration of diquafosol sodium 3% compared to sodium hyaluronate 0.1%

Participants will receive diquafosol sodium 3% or sodium hyaluronate 0.1% for 4 weeks before the cataract surgery and 21 days after the surgery.

The steps of the research examination are as follows:

A) History

* Comorbid dry eye disease and screening exclusion criteria (history of smoking, previous medical history, history of hypertension, history of diabetes mellitus, history of routine medication and history of recent surgery)
* Ocular Surface Disease Index (OSDI) Questionnaire

B) Physical Examination

The examination is carried out with sufficient lighting, to see if the patient's eye has other eye surface disorders that can affect dry eye syndrome. Examination of disorders of the surface of the eyeball is carried out by inspection to see the patient's ability to blink, the eyelids, eyelashes and interpalpebral surface, performing an examination by lifting the upper upper eyelid superiorly, examination by pulling the eyelid to see if the eyelid looks drooping and checking In the fornix of the eye, emphasis is placed on the expression of the meibomian glands. The existence of a positive examination, describes the patient has a disorder of the eyeball surface. This examination determines whether the patient can undergo cataract surgery for research.

C) Supporting Examination

- Contrast sensitivity using the Pelli-Robson diagram, keratograph, HOA, tear osmolarity, MMP-9, corneal sensitivity, tear break up time, fluorescein break up pattern.

This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Cataract patients who will undergo phacoemulsification procedures and intraocular lens (IOL) implants
2. Patients with dry eye disease
3. Patients are willing to participate in the study and fill out informed consent

Exclusion Criteria:

1. Subjects with lacrimal gland or eyelid disorders (ptosis, blepharospasm, lagophthalmos, entropion, ectropion, and blepharitis)
2. There are complications after cataract surgery
3. Patients with a history of using topical medications / eye drops that are used routinely
4. History of eye surgery in the last 6 months
5. Serious ocular surface disorders (Sjögren syndrome, pemphigoid, chemical trauma)
6. Using regular medication that trigger dry eye conditions (eg antihistamines, antidepressants, decongestants, anticholinergics) / allergy to diquafosol drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
OSDI questionnaire score | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients subjectively with OSDI questionnaire. The OSDI score results will be assessed. Lower scores mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Tear break up time value | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients objectively by examining the value of tear break up time. Higher value in tear break up time mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Fluorescein break up pattern | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients objectively by examining the fluorescein break up pattern. The fluorescein break up pattern results will be categorized and analyzed descriptively.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Corneal sensibility using Cochet Bonnet esthesiometer | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients objectively by examining the value of corneal sensibility using cochet bonnet esthesiometer. Any changes to the value will be assessed. Higher value mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Tear osmolarity using TearLab device | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients subjectively objectively by examining the value of tear osmolarity using TearLab device. Lower value mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Higher Order Aberrations (HOA) value using oculyzer device | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients objectively by examining the value of Higher Order Aberrations (HOA) using oculyzer device to assess the corneal aberrations. Lower value mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Contrast sensitivity value using Pelli-Robson Contrast Sensitivity Chart | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients objectively by examining the value of contrast sensitivity using Pelli-Robson Contrast Sensitivity Chart. Higher value mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Matrix metalloproteinase-9 value using Human MMP-9 ELISA Kit | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients objectively by examining the value of matrix metalloproteinase-9 using Human MMP-9 ELISA Kit. Lower value mean a better outcome.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.
Keratograph device to assess tear meniscus height, noninvasive keratograph tear break up time (NIKBUT), and redness | 4 months
  This study will evaluate differences in the use of diquafosol sodium 3% and sodium hyaluronate 0.1% in improving dry eye disease signs and symptoms in patients subjectively objectively by examining the patients using keratograph device to assess the tear meniscus height, noninvasive keratograph tear break up time (NIKBUT), and redness. The results will be categorized and analyzed descriptively.
  This examination will be carried out 4 times: on the first day before the research series, four weeks after giving therapy before cataract surgery, 21 days after cataract surgery, and 90 days after cataract surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia